CLINICAL TRIAL: NCT06201143
Title: The Effect of kınesıologıcal tapıng, mobılızatıon and breathıng exercıse on paın and Comfort After Caesarea
Acronym: Caesarea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Şırnak Üniversitesi (Other)
Responsible Party: Principal Investigator, Kübra Akcan, lecturer, Şırnak Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SirnakU
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Nurse; Cesarean Section; Postpartum Comfort
Keywords: pain; nurse; kinesiology taping; pospartum comfort; breathing exercise; mobilization
MeSH Terms: conditions — Pain | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP (Experimental): Breathing exercise and mobilization training will be given in the patient's room during the preoperative period. Each training is planned to last approximately 20 minutes. Respiratory and mobilization training for patients during training techniques will be taught in practice, they will be shown how to mark the breathing exercise and mobilization tracking chart, and their questions will be answered.
  Individuals in this group will be given breathing exercise and mobilization training. VAS form will be filled in at the 10th, 24th, 48th and 72nd hours of postpartum. The patient's total mobilization time and the number of breathing exercises will be recorded. The postpartum comfort scale will be filled in at the 10th and 72nd hours.
  Interventions: Other: BREATHING EXERCISE AND MOBILIZATION TRAINING
- KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP (Experimental): Participants in this group will be given kinesiology taping, breathing exercise and mobilization training. Kinesiological taping will be done at the 10th hour postoperatively. The VAS form will be filled out at the 10th, 24th, 48th and 72nd postoperative hour. The patient's total mobilization time and the number of breathing exercises will be recorded. The postpartum comfort scale will be filled in at the 10th and 72nd hours.
  Interventions: Other: BREATHING EXERCISE AND MOBILIZATION TRAINING; Other: KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING
- CONTROL GROUP (No Intervention): No intervention will be made to individuals participating in this group. The VAS form will be filled out at the 10th, 24th, 48th and 72nd postoperative hour. The patient's total mobilization time and the number of breathing exercises will be recorded. The postpartum comfort scale will be filled in at the 10th and 72nd hours.

INTERVENTIONS:
Other: BREATHING EXERCISE AND MOBILIZATION TRAINING — After cesarean mobilization and breathing exercise training, the number of breathing exercises performed and the duration of mobilization will be recorded. Thus, the effectiveness of the training will be examined in detail.
  Arms: BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP; KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP
Other: KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING — It will be the first study to use kinesiotaping, breathing exercise and mobilization training together.
  Arms: KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP

SUMMARY:
No study has been found in which kinesiology taping, mobilization and breathing exercises were used regarding postoperative pain and postpartum comfort after cesarean section. This study aims to determine the effects of kinesiology taping, mobilization and breathing exercise on post-cesarean section pain and postpartum comfort.

The study will be conducted with three groups, two intervention groups and one control group. It has been calculated that a minimum of 33 people in each group and 99 people in total will be sufficient. Anticipating the possibility of data loss in the study, it was planned to include 15% more patients (n = 114).

Research Questions Is there a difference in terms of pain between the groups that received kinesiology taping, mobilization training and breathing exercises after cesarean section and those that did not? Is there a difference in postpartum comfort level between the groups that received kinesiology taping, mobilization training and breathing exercises after cesarean section and those that did not? Is there a difference in terms of pain between groups with and without post-cesarean mobilization training and breathing exercise? Is there a difference in postpartum comfort level between groups with and without post-cesarean mobilization training and breathing exercise?

DETAILED DESCRIPTION:
This study was designed with quantitative research method. Randomized controlled experimental design of quantitative research will be used in this study. It will be conducted with women who are in the postoperative period after cesarean section and who volunteer to participate in the research. The population of the research consists of women who were admitted to Şırnak State Hospital gynecology clinic and had a cesarean section in the last year. The sample size and power calculation required for the study were calculated with the G*Power Ver.3.1.9.2 program. It was calculated that 99 people would be sufficient. Anticipating the possibility of data loss in the study, it was planned to include 15% more patients (n = 114). Thus, the study was planned to be conducted with 38 participants in each group and 114 participants in total. This research will be a randomized controlled trial. Randomization of the groups will be done in a simple random manner using the website www.random.org. The study will be conducted with three groups, two intervention groups and one control group. Participants will be placed into groups according to the randomization list. Mothers who meet the sample selection criteria and agree to participate in the research will be included in the research. As a data collection tool; Introductory information form, Mobilization and Respiratory Exercise Follow-up Chart, Visual Analogue Scale =VAS and Postpartum Comfort Scale will be used.

COLLECTION OF DATA BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP Pregnant women who are admitted to the gynecology ward for cesarean section, who agree to participate in the study and who meet the sample selection criteria will be assigned to the application group according to the randomization list. Pregnant women will be interviewed before the cesarean section, an explanation will be given about the purpose of the research, its content and the methods to be applied, and an informed consent form will be obtained verbally and in writing. Pregnant women will fill in the sections of the introductory information form questioning sociodemographic and obstetric characteristics through face-to-face interviews. Mothers will be asked to sleep in different rooms to prevent interaction with each other.

Breathing exercise and mobilization training will be given in the patient's room during the preoperative period. Each training is planned to last approximately 20 minutes. During the training, patients will be taught breathing and mobilization techniques in practice, will be shown how to mark the breathing exercise and mobilization tracking chart, and their questions will be answered.

The patient will be informed about techniques and points to consider regarding sitting on the edge of the bed, standing up on the edge of the bed, and walking in the patient room, as well as the time he/she will spend out of bed on the day of surgery and the first and subsequent days after surgery.

The patient will be informed that he or she will need to be mobilized out of bed for 2 hours on postoperative day 0 and for 6 hours on postoperative day 1 and thereafter. Six hours after the surgery, the patient's first mobilization will be performed by the researcher. The patient will be mobilized by planning the second and third mobilization at four-hour intervals. Outside of planned mobilization hours, patients will be informed about mobilization as long as they feel well.

The patient will be told that breathing exercises should be done on the day of surgery, on the first and second days after surgery, when the patient is awake and able to move freely, 5 sets of 10 repetitions a day. Since pursed lip exercise is used in studies conducted after abdominal surgery in the literature, pursed lip exercise will be taught in breathing exercise training.

In order to increase lung expansion, the patient will be placed in the Fowler position and instructed to take a slow deep breath through his nose, hold it in for two or three seconds, and slowly purse his lips at the time of expiration. In line with the literature, breathing exercises will be required to be performed 5 sets of 10 repetitions a day.

The patient will be taught to wait 1-2 seconds after each breath. A breathing exercise and mobilization training brochure prepared in line with the literature will be given to the patients.

VAS will be filled at the 10th postoperative hour. Simultaneously with the kinesiology taping + breathing exercise and mobilization training group, VAS will be filled in again 45 minutes after the first VAS evaluation.

VAS measurements will be repeated at the 24th, 48th and 72nd hours postoperatively.

The first measurement of the postpartum comfort scale will be completed at the 10th postoperative hour, and the second measurement will be completed at the 72nd postoperative hour.

The mother will be asked to record the times of gas and stool passage and these will be recorded in accordance with the patient's statement.

KINESIOLOGICAL TAPING + BREATHING EXERCISE AND MOBILIZATION TRAINING GROUP; Pregnant women who are admitted to the gynecology ward for cesarean section and who meet the research criteria will be interviewed before the cesarean section, an explanation will be given about the purpose of the research, its content and the methods to be applied, and verbal and written informed consent forms will be obtained from those who wish to participate in the study. Pregnant women will fill in the sections of the introductory information form questioning their sociodemographic and past obstetric characteristics through face-to-face interviews.

Breathing exercise and mobilization training will be given in the patient's room during the preoperative period. Each training is planned to last approximately 20 minutes. During the training, patients will be taught breathing and mobilization techniques in practice, will be shown how to mark the breathing exercise and mobilization tracking chart, and their questions will be answered.

The patient will be informed about techniques and points to consider regarding sitting on the edge of the bed, standing up on the edge of the bed, and walking in the patient room, as well as the time he/she will spend out of bed on the day of surgery and the first and subsequent days after surgery.

The patient will be informed that he or she must provide out-of-bed mobilization for 2 hours on postoperative day 0 and 6 hours on postoperative day 1 and thereafter.

On the day of surgery, the first mobilization of the patient will be performed by the researcher six hours after the surgery. The patient will be mobilized by planning the second and third mobilization at four-hour intervals. Outside of planned mobilization hours, patients will be informed about mobilization as long as they feel well.

The patient will be told that breathing exercises should be done on the day of surgery, on the first and second days after surgery, when the patient is awake and able to move freely, 5 sets of 10 repetitions a day.

In line with the literature, preoperative breathing exercise and mobilization training booklet will be given to patients.

What happens in the 10th postoperative hour for kinesiology taping: In the first 10 hours after the surgery, hypotension due to bleeding during the surgery and the effect of anesthesia and the resulting weakness, headache due to dural puncture, dizziness, nausea and vomiting, complaints of low back pain are frequently observed, numbness in the extremities is observed in women, Kinesiology taping will be started postoperatively in order to remain cognitively under the influence of anesthesia and to effectively apply measurement tools and applications. Kinesiology tape comes in blue, cream, pink and black colors. The color choice of the band is left to the patients' preference. I tape will be adhered around the incision area with the web cutting technique, leaving the incision area open, using the space conservation technique, without applying tension to the starting and ending points. After application, the tape will be adhered to by hand movements.

In order to facilitate the patients' gas and stool passage, the I band will be turned into a Y band, and four bands, two on the right and left, will be attached around the belly with circulatory/lymphatic correction technique with 25% tension on the tails, without tension at the starting point.

In line with the literature, VAS will be filled in immediately before kinesiology tape applications (at 10 hours postoperatively) and 45 minutes after the application in order to observe acute pain.

VAS measurements will be repeated at 24, 48 and 72 hours postoperatively. The first measurement of the postpartum comfort scale will be completed at the 10th postoperative hour, and the second measurement will be completed at the 72nd postoperative hour.

After completing the questionnaires, the tapes will be removed by the researcher using baby oil.

During the study, patients' questions will be answered and counseling will be provided during face-to-face meetings.

The mother will be asked to record the times of gas and stool passage and these will be recorded in accordance with the patient's statement.

The structured information form, scales and kinesiology tape application steps will be applied by the researcher who has completed the Kinesiotaping 1-2 Certificate Course.

CONTROL GROUP; Pregnant women who are admitted to the gynecology ward for cesarean section, who agree to participate in the study and who meet the sample selection criteria will be assigned to the application group according to the randomization list. Pregnant women will be interviewed before the cesarean section, an explanation will be given about the purpose of the research, its content and the methods to be applied, and an informed consent form will be obtained verbally and in writing. Pregnant women will fill in the sections of the introductory information form questioning their sociodemographic and past obstetric characteristics through face-to-face interviews. Mothers will be asked to sleep in different rooms to prevent interaction with each other.

ELIGIBILITY:
Inclusion Criteria:

Must be in the 18-45 age group 37-40. There should be a cesarean section during the gestational week. Should not have a chronic disease Must not have a dermatological disease

Exclusion Criteria:

Deep vein thrombosis, open wound or skin irritation, etc.), Participants whose babies were taken to the neonatal intensive care unit

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Skala | It will be filled in at the 10th, 24th, 48th and 72nd postoperative hours.
  "Participants obtained a response when they rated 0 or 10 performance states on a scale ranging from 0 (best outcome) to 10 (worst outcome).

IPD SHARING:
Plan to Share IPD: No